CLINICAL TRIAL: NCT00217841
Title: A Multi Centre, Double-Blind, Randomised, Placebo Controlled Prospective Study on the Safety and Efficacy of Aurograb in Patients With Severe, Deep-Seated Staphylococcal Infections Receiving Vancomycin
Brief Title: Aurograb and Vancomycin in MRSA Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NeuTec Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: NTP/Aurograb/003
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Staphylococcal Infections
Keywords: MRSA
MeSH Terms: conditions — Staphylococcal Infections

INTERVENTIONS:
Drug: Aurograb

SUMMARY:
The study hypothesis is that the addition of Aurograb to standard vancomycin therapy will improve outcome in MRSA infection.

DETAILED DESCRIPTION:
The Primary Objective will be to determine whether the overall response (clinical and bacterial) to Aurograb® (1mg/kg i.v. b.d.) plus vancomycin is greater than the overall response to placebo plus vancomycin, in adult hospitalised patients with severe, deep-seated staphylococcal infections, particularly MRSA infections, being treated with vancomycin.

Secondary Objectives will be:

1. To further determine efficacy, comparing Aurograb versus placebo, regarding:

   * attributable mortality
   * overall mortality
   * clinical response
   * bacterial response ie eradication or persistence of the infection
   * rates of clinical resistance to vancomycin.
2. To compare the safety profile of treatment with Aurograb® (1mg/kg b.d.) plus vancomycin versus placebo plus vancomycin in adult hospitalised patients with deep-seated staphylococcal infections.
3. To extend the data base on pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

All patients will have to satisfy the following inclusion criteria to enter the study:

* Hospitalised adult patients (18 years or over) with severe, deep-seated staphylococcal infection being treated with vancomycin, this diagnosis being based on clinical signs and symptoms appropriate to the site of infection (as detailed under subsets, Section 4.6) plus a positive culture or Gram stain showing Gram positive cocci in clusters (not chains) from one or more of the following clinically significant sites:

  i. a blood culture ii. a lower respiratory tract specimen eg sputum or BAL iii. pleural fluid iv. intra-abdominal fluid or tissue v. urine (in patients with renal sepsis or complicated urinary tract infections)
* The study drug must be started while there is clinical evidence of active infection (usually within 24 hours of starting vancomycin, although longer delays are acceptable if the patient is still clinically septic and culture positive within 24 hours of starting study drug).
* Recruitment may be initiated on the basis of a Gram stain but, for the patient to be eligible to continue in the study, staphylococcal sepsis must subsequently be confirmed by culture.
* The positive specimen must be from a clinically significant specimen taken within 2 days of starting the study drug.
* Patients must be on i.v. vancomycin as the sole systemic antibiotic for the first 3 days of the study.
* Patients must have sufficient venous access to permit administration of study drug and monitoring of safety variables
* Written informed consent must be obtained for participation in the study.

Exclusion Criteria:

Patients fulfilling the following criteria will not enter the study:

* Prior Antibiotic Usage: Patients who have received (within 48 hours of study entry) a systemic anti-staphylococcal antibiotic other than vancomycin for longer than 24 hours, unless the patient was considered to have failed that regime ie a documented treatment failure (ie 3 days' treatment and not responding) or the Staphylococcus is resistant to the antibiotic in vitro (e.g. the patient is initially treated with flucloxacillin but the isolate subsequently identified as resistant) - in such cases the antibiotic must be changed to vancomycin to enter the study.
* Concomitant Antibiotics: usage of concomitant antibiotic except as allowed by the protocol (see Section 5.3)
* Patients with devices infected with S. aureus, including implants and catheters, which cannot be removed
* Patients known to have AIDS, who have a CD4 cell count < 200 cells/mm3
* Patients with staphylococcal endocarditis, mediastinitis, meningitis, osteomyelitis and/or joint infections.
* Asymptomatic carriers of MRSA - such patients must be clinically septic due to the MRSA
* Patients with methicillin-sensitive CNS (MSSE)
* Patients with methicillin-resistant CNS (MRSE) unless they are clinically significant blood culture isolates, as indicated by two blood cultures (taken from two different sites) growing the same CNS in a clinically septic patient in whom there is no other significant pathogen responsible for the sepsis
* Females who have a positive pregnancy test
* Patients who have a known allergy to any constituent of Aurograb® (i.e. hypersensitivity to antibody, nickel, urea or arginine)
* Patients who have received an unlicensed drug within three months prior to the study
* Patients with a concomitant medical condition, in whom, in the opinion of the Investigator, participation may create an unacceptable risk for the patient
* Patients considered inappropriate for enrolment in this study by the Investigator for any other reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2004-01; Study Completion 2006-03

PRIMARY OUTCOMES:
The response to Aurograb® (1mg/kg i.v. b.d.) plus vancomycin is greater than the overall response to placebo plus vancomycin,in patients with severe, deep-seated staphylococcal infections.

SECONDARY OUTCOMES:
attributable mortality
overall mortality
clinical response
bacterial response
rates of clinical resistance to vancomycin.
To extend the data base on pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Wilcox, MD, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- Mark Wilcox, Leeds, England, United Kingdom

REFERENCES:
- [Background] Burnie JP, Matthews RC, Carter T, Beaulieu E, Donohoe M, Chapman C, Williamson P, Hodgetts SJ. Identification of an immunodominant ABC transporter in methicillin-resistant Staphylococcus aureus infections. Infect Immun. 2000 Jun;68(6):3200-9. doi: 10.1128/IAI.68.6.3200-3209.2000. PMID 10816464